CLINICAL TRIAL: NCT03222635
Title: Endoscopic Management of Patients With High Risk T1a and T1b N0M0 Esophageal Adenocarcinoma: a Prospective Multicenter Registry.
Brief Title: Prospective Endoscopic Follow-up of Patients With Submucosal and High Risk Mucosal Esophageal Adenocarcinoma
Acronym: PREFER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Jacques J.G.H.M. Bergman, Professor of Gastrointestinal Endoscopy, Amsterdam UMC, location VUmc
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL6116501817
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Submucosal Esophageal Adenocarcinoma; Barrett Esophagus; High-risk Mucosal Esophageal Adenocarcinoma
Keywords: Barrett's esophagus; Submucosal esophageal adenocarcinoma; Endoscopic treatment; Endoscopic follow-up; High-risk mucosal esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Upon achieving the designated sample size of 141 patients of the original PREFER-trial, the enrolment of further patients diagnosed with T1b N0M0 EAC and treated endoscopically will be continued as a registration cohort (no sample size) within the same study database.
  The high-risk T1a group will also continue as a registration cohort, since there is no available data yet to calculate a reliable sample size with. The high-risk T1a patient group will be analysed separately from the T1b patient group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic follow-up (Experimental): Patients treated with endoscopic resection (ER) for a submucosal or high-risk mucosal esophageal adenocarcinoma without lymphnode- or distant metastases (N0M0) will undergo endoscopic follow-up.
  Interventions: Procedure: Endoscopic follow-up

INTERVENTIONS:
Procedure: Endoscopic follow-up — Endoscopic follow-up by means of regular upper endoscopies and endoscopic ultrasounds

SUMMARY:
Aim of this prospective multicenter study is to evaluate the safety of an endoscopic follow-up strategy in patients treated with endoscopic resection (ER) for submucosal or high-risk mucosal esophageal adenocarcinoma (T1bN0M0 or HR T1aN0M0 EAC).

DETAILED DESCRIPTION:
Traditionally, the risk of lymph node metastasis associated with submucosal EAC was considered too high to offer patients endoscopic follow-up. Only in elderly patients with comorbidity, more often an endoscopic protocol is selected. However, the risk of lymph node metastasis associated with submucosal EAC is mainly based on surgical series. Recently a number of studies, which included patients treated endoscopically, were published indicating that the risk of lymph node metastasis may be much lower than generally assumed (1-5). Therefore, a less invasive and organ preserving approach may not only be an option in the frail and elderly, but for all patients with submucosal EAC's.

Yet, no data exists on the risk of lymph node metastasis in high risk T1a EAC. The risk is assumed to be lower than for EACs invading into the submucosal layer. However, a recent retrospective analysis from our own research group shows that this risk may be higher than previously assumed (6). In this nationwide retrospective study, we analyzed lymph node metastasis rates and EAC related mortality rates concerning patients with high risk T1a, low risk T1b or high risk T1b EAC who received endoscopic treatment. The study was performed in 9 Barrett Expert Centers in the Netherlands (2008-2019). 120 patients were included in the analysis, and results showed the highest lymph node metastasis risk in the high risk T1a patient group.

Aim of this multicenter study is to prospectively evaluate the safety of endoscopic follow-up in patients treated by endoscopic resection for submucosal (T1bN0M0) and high risk mucosal (T1aN0M0) EAC.

High-resolution upper endoscopy with white-light endoscopy and narrow-band imaging supplemented with an EUS are performed every three months during the first two years after ER. After 1 year, a CT-thorax/abdomen will be performed to check for distant metastasis. During the third and fourth year of follow-up, EUS and upper endoscopy are performed every six months. From the fifth year on, EUS and upper endoscopy are performed annually.

ELIGIBILITY:
Inclusion Criteria:

* Patients with submucosal or high-risk mucosal EAC diagnosed in an ER specimen, by an expert gastrointestinal (GI) pathologists.
* Signed informed consent.

Exclusion Criteria:

* Prior history of high-risk mucosal or ≥T1sm.
* Synchronous esophageal squamous cell carcinoma.
* Suspicion on lymph node metastasis or distant metastasis on EUS, ultrasound of the neck or CT-thorax-abdomen performed six weeks after ER during baseline measurement.
* Tumor-positive deep resection margin (R1) in ER specimen.
* Patients unable to give signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2028-07-25 (Estimated); Study Completion 2028-07-25 (Estimated)

PRIMARY OUTCOMES:
5-year disease-specific mortality/survival (descriptive statistics in SPSS, percentages, survival analysis) | 5 years
  Disease specific mortality is decribed as mortality directly linked to the esophageal adenocarcinoma (i.e., metastasized EAC, metastasized disease with a simultaneously primary cancer present and it cannot be ruled out (based on histology) that the metastases are related to the other primary cancer, death due to complications of the endoscopic procedure, death due to complications after surgery or CRT, no clear cause of death in patients who have metastases or untreated local recurrence). If patients are diagnosed with distant metastases, and subsequently die of a non-tumor related cause, patients will still be documented as tumor-related death. Will be measured in number of patients and percentages. Survival analysis using Kaplan Meier will be performed.
Overall survival (descriptive statistics in SPSS, percentages, survival analysis) | 5 years
  Overall survival of study population (tumor-related + non-tumor-related deaths). Measured in numbers and percentages, survival analysis (KM).

SECONDARY OUTCOMES:
Lymph node metastasis, confirmed by cytology and/or histology (descriptive statistics in SPSS, number of patients (%)) | 5 years
  Confirmed by cytology and/or histology by performing FNA during EUS or biopsies.
Local recurrence eligible for endoscopic therapy (descriptive statistics in SPSS, number of patients (%)) | 5 years
  In case a local recurrence is found during FU endoscopy, histopathology have to show if it is recurrent cancer.
Local recurrence requiring surgical therapy (descriptive statistics in SPSS, number of patients (%)) | 5 years
  In case a local cancer recurrence is not amendable for endoscopic re-treatment, for example due to extensive disease or fibrosis, a patient will be referred for surgery if possible.
Distant metastasis, histologically proven (descriptive statistics in SPSS, number of patients (%)) | 5 years
  Primary tumor of distant metastasis should be histopathologically evalueted by taking biopsies.
Quality of life during follow-up endoscopies (questionnaires) | 5 years
  Quality of life is assessed by using questionnaires on set time points during the whole study.

CONTACTS AND LOCATIONS:
Overall Officials: J. J. Bergman, MD, PhD, Principal Investigator — Amsterdam UMC; R. E. Pouw, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (20):
- Westmead hospital, Sydney, Australia
- Belgium (4):
  - CUB Hôpital Erasme, Brussels
  - AZ Maria Middelares Ghent, Ghent
  - UZ Leuven, Leuven
  - AZ Delta Roeselare, Roeselare
- Germany (4):
  - Universitätsklinikum Augsburg, Augsburg
  - EVK Duesseldorf, Düsseldorf
  - MRI TUM, Münich
  - Barmherzige Brüder Regensburg, Regensburg
- Netherlands (8):
  - Amsterdam UMC, Amsterdam
  - Catharina Hospital, Eindhoven
  - University Medical Center Groningen, Groningen
  - St. Antonius Hospital, Nieuwegein
  - Radboudumc, Nijmegen
  - Erasmus MC - University Medical Center, Rotterdam
  - Haga Medical Center, The Hague
  - Isala Clinics, Zwolle
- Hirslanden private hospital group, Zurich, Switzerland
- United Kingdom (2):
  - University College London Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez Herrero L, Pouw RE, van Vilsteren FG, ten Kate FJ, Visser M, van Berge Henegouwen MI, Weusten BL, Bergman JJ. Risk of lymph node metastasis associated with deeper invasion by early adenocarcinoma of the esophagus and cardia: study based on endoscopic resection specimens. Endoscopy. 2010 Dec;42(12):1030-6. doi: 10.1055/s-0030-1255858. Epub 2010 Oct 19. PMID 20960392
- [Background] Scholvinck D, Kunzli H, Meijer S, Seldenrijk K, van Berge Henegouwen M, Bergman J, Weusten B. Management of patients with T1b esophageal adenocarcinoma: a retrospective cohort study on patient management and risk of metastatic disease. Surg Endosc. 2016 Sep;30(9):4102-13. doi: 10.1007/s00464-016-5071-y. Epub 2016 Jun 29. PMID 27357927
- [Background] Manner H, May A, Pech O, Gossner L, Rabenstein T, Gunter E, Vieth M, Stolte M, Ell C. Early Barrett's carcinoma with "low-risk" submucosal invasion: long-term results of endoscopic resection with a curative intent. Am J Gastroenterol. 2008 Oct;103(10):2589-97. doi: 10.1111/j.1572-0241.2008.02083.x. Epub 2008 Sep 10. PMID 18785950
- [Background] Manner H, Pech O, Heldmann Y, May A, Pohl J, Behrens A, Gossner L, Stolte M, Vieth M, Ell C. Efficacy, safety, and long-term results of endoscopic treatment for early stage adenocarcinoma of the esophagus with low-risk sm1 invasion. Clin Gastroenterol Hepatol. 2013 Jun;11(6):630-5; quiz e45. doi: 10.1016/j.cgh.2012.12.040. Epub 2013 Jan 26. PMID 23357492
- [Background] Manner H, Pech O, Heldmann Y, May A, Pauthner M, Lorenz D, Fisseler-Eckhoff A, Stolte M, Vieth M, Ell C. The frequency of lymph node metastasis in early-stage adenocarcinoma of the esophagus with incipient submucosal invasion (pT1b sm1) depending on histological risk patterns. Surg Endosc. 2015 Jul;29(7):1888-96. doi: 10.1007/s00464-014-3881-3. Epub 2014 Oct 8. PMID 25294553
- [Background] Nieuwenhuis EA, van Munster SN, Meijer SL, Brosens LAA, Jansen M, Weusten BLAM, Alvarez Herrero L, Alkhalaf A, Schenk E, Schoon EJ, Curvers WL, Koch AD, van de Ven SEM, Verheij EPD, Nagengast WB, Westerhof J, Houben MHMG, Tang T, Bergman JJGHM, Pouw RE; Dutch Barrett Expert Centers. Analysis of metastases rates during follow-up after endoscopic resection of early "high-risk" esophageal adenocarcinoma. Gastrointest Endosc. 2022 Aug;96(2):237-247.e3. doi: 10.1016/j.gie.2022.03.005. Epub 2022 Mar 12. PMID 35288149